CLINICAL TRIAL: NCT03273361
Title: Desk-Compatible Elliptical Device: Feasibility Evaluation
Brief Title: Desk Cycling Work Performance Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Liza Rovniak, Associate Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00001535
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Physical Activity; Overweight
MeSH Terms: conditions — Obesity; Motor Activity; Overweight

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects were randomly assigned to a pedaling sequence based on the Graeco Latin squares design. They were blinded regarding which pedaling sequence they were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Seated (Experimental): Participants completed work tasks while seated.
  Interventions: Behavioral: Compact Cycling Device
- Low Intensity Pedaling (Experimental): Participants completed work tasks while pedaling at a low intensity.
  Interventions: Behavioral: Compact Cycling Device
- Low-Moderate Intensity Pedaling (Experimental): Participants completed work tasks while pedaling at a low-moderate intensity.
  Interventions: Behavioral: Compact Cycling Device

INTERVENTIONS:
Behavioral: Compact Cycling Device — Participants pedaled a compact cycling device while simultaneously working at a desk.

SUMMARY:
This lab study is evaluating the feasibility of accomplishing productive office work while simultaneously pedaling a compact desk-based cycling device.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Ability to type without looking at the keyboard
* Native English speaker
* Normal hearing
* Spend 6 or more hours per day sitting
* Less than 150 minutes of physical activity per week

Exclusion Criteria:

* Positive response on the Physical Activity Readiness Questionnaire indicating that low intensity pedaling could present safety risks
* Pregnancy
* Body mass index less than 18 or greater than 35

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Typing task | 5 minutes
  Participants completed a computerized typing task

SECONDARY OUTCOMES:
Reading task | 5 minutes
  Participants read a brief passage and answered questions to assess reading comprehension.
Logic Reasoning and Phone Task | 5 minutes
  Participants completed logical reasoning questions while answering a simulated phone call.

CONTACTS AND LOCATIONS:
Overall Officials: Liza Rovniak, PhD, MPH, Principal Investigator — Pennsylvania State University College of Medicine; Andris Freivalds, PhD, Study Director — Penn State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rovniak LS, Cho J, Freivalds A, Kong L, DE Araujo-Greecher M, Bopp M, Sciamanna CN, Rothrock L. Effects of Desk Pedaling Work Rate on Concurrent Work Performance among Physically Inactive Adults: A Randomized Experiment. Med Sci Sports Exerc. 2023 Jan 1;55(1):20-31. doi: 10.1249/MSS.0000000000003026. Epub 2022 Aug 16. PMID 35977110